CLINICAL TRIAL: NCT05661565
Title: Correlation of Insulin Resistance With Hormonal and Ovarian Morphological Characteristics in Patients With Polycystic Ovarian Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fatma Fathy Hafez Ismail, principle investigator, NewGiza University
Other Study IDs: 0000000
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Study the Relationship Between Insulin Resistance With Hormonal and Ovarian Morphological Characteristics in Patients With Polycystic Ovarian Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — We try to find an association between insulin resistance with ovarian hormonal and morphological characteristics in patients with polycystic ovarian syndrome

SUMMARY:
We designed a study to determine if ovarian volume (OV) and/or follicle number (FN) are independently associated with abnormal metabolic findings in women diagnosed with PCOS. We hypothesized that ovarian morphology but not follicle number would be associated with a significantly higher odds of hyperinsulinemia among women with PCOS.

ELIGIBILITY:
Inclusion Criteria:

A-patients met the Rotterdam criteria of PCO with two out of three of the following:

1. oligo-or-anovulation
2. clinical and/or biochemical hyperandrogenism
3. the presence of 10 or more antral follicles in one ovary and/or a maximum ovarian volume > 10cc B-reproductive age group (16:45 years) C-BMI <40

Exclusion Criteria:

A-age >40 years B-BMI>40 C-previous ovarian surgery D-chronic medical disorders [DM , HTN , ...]

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Women with PCOS attending the outpatient clinic in Kasr Alainy Hospital in the reproductive age group (20:40 years)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between the ovarian volume and Insulin resistance | January 2023- June 2023
Correlation between the antral follicular count and insulin resistance | January 2023- June 2023

SECONDARY OUTCOMES:
Correlation between anti-mullerian hormone values and insulin resistance | January 2023- June 2023
Correlation between FSH values and insulin resistance | January 2023- June 2023
Correlation between LH values and insulin resistance | January 2023- June 2023
Correlation between body mass index and insulin resistance | January 2023- June 2023
Correlation between hirsutism and insulin resistance | January 2023- June 2023

IPD SHARING:
Plan to Share IPD: Undecided